CLINICAL TRIAL: NCT05027035
Title: Diaphragm Paralysis: Surgery or Mechanical Ventialion
Acronym: PARASOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Peter Wijkstra, Prof. Dr. P.J. Wijkstra, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 80-87700-98-22188
Record Dates: First submitted 2021-08-01; First posted 2021-08-30 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diaphragm Paralysis
Keywords: mechanical ventilation; surgical plication of the diaphragm
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Intervention Model Description: open-label, multi center, intervention pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical plication (Active Comparator): Surgical plication of the diaphragm
  Interventions: Other: surgical plication" or "nocturnal non-invasive ventilation
- Mechanical ventilation (Active Comparator): Non-invasive ventiatilatory support while on the waiting list for surgical plication
  Interventions: Other: surgical plication" or "nocturnal non-invasive ventilation

INTERVENTIONS:
Other: surgical plication" or "nocturnal non-invasive ventilation — 10 participants for surgical plication and 10 participants for nocturnal non-invasive ventilation.

SUMMARY:
Summary Rationale: The diaphragm is a dome-shaped muscle which separates the thoracic cavity from the abdomen. In patients with diaphragm paralysis the treatment (surgery versus non-invasive ventilation) is based on physician preference, not sound scientific evidence. Clearly studies are needed to guide a scientific decision making.

Objective: In this pilot study the we want to know the clinical relevant effect of both therapies on EQ-5D_5L, the latter being the primary outcome. Finally, it will show the investigators the costs of both therapies form a societal perspective.

Study design: open-label, multi center intervention pilot study Study population: 20 participants >18 year and diagnosed with a unilateral diaphragm paralysis resulting from phrenic nerve injury.

Intervention: 10 participants for surgical plication and 10 participants for nocturnal non-invasive ventilation while on the wating list for surgical plication.

Main study parameters/endpoints:

The goal of the pilot study is to describe the effect of both plication and NIV on the endpoints of the intended efficiency study. The intended primary endpoint is quality of life as measured by the EQ-5D-5L questionnaire. Secondary endpoints are; the Medical Research Council (MRC) dyspnoea scale, the Diaphragmatic Paralysis Questionnaire, Borg dyspnoea score, 6 minute walk test, spirometry in both sitting and supine position, a polysomnography and transcutaneous measurement of carbon dioxide an oxygen saturation at night.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

The diaphragm is a dome-shaped muscle which separates the thoracic cavity from the abdomen. It is the most important muscle of respiration innervated by the phrenic nerves. While many diseases might interfere with its function (1), in the intended study the investigators will focus on diaphragm paralysis due to phrenic nerve injury. Two types of diaphragm paralysis can be distinguished: unilateral and bilateral. Patients with unilateral paralysis perceive exertional dyspnea, have an impaired exercise capacity and orthopnea.(2) Patients with a bilateral paralysis usually have more symptoms and might even develop respiratory failure. (3) In addition, all patients with a diaphragm paralysis may have poor sleep quality, as the diaphragm is the only active respiratory muscle during REM sleep. (4) Currently, two treatment approaches for patients with diaphragm paralysis are used in clinical practice: surgical diaphragm plication and nocturnal non-invasive ventilation (NIV). Plication is a minimal invasive surgical procedure that aims to stiffen the diaphragm and such limits dysfunctional (paradoxical movement) excursions of the paralytic diaphragm. The procedure is performed in ±70 patients per year in the Netherlands. NIV is a non-invasive mode of positive pressure ventilatory assistance; through a facial mask the ventilator supports patient breathing effort. Patients with diaphragm paralysis use their ventilator mainly during night time, to improve quality of sleep and such to reduce day time symptoms. In the Netherlands, home mechanical ventilation is very well organized, as care is delivered by only 4 specialized centers. NIV for diaphragm paralysis is started in around 50 patients yearly.

Currently, both plication and nocturnal NIV appear beneficial and both options are covered by health care insurance. However, it is unknown which intervention is most beneficial from a patient perspective. For instance, comparison on patient relevant outcome measures and complications between these treatment approaches is unknown. In addition, patients with diaphragm paralysis may develop severe symptoms, limiting daily activities including ability to perform their professional work. To assess the overall impact of this a detailed cost analysis is necessary to compare both treatments from a societal perspective. A solid cost effectiveness / cost utility study will reveal which therapy is the best option from a societal perspective.

This pilot study will be set up as an intervention study.To know what clinical effect of both therapies is relevant the EQ-5D-5L is used. It is unknown whether there is a significant difference on the outcome between both therapies. A search in trial registries did not reveal any study with similar research questions. Based on the outcomes of this preparatory study a power analysis can be performed for the seminal study. Due to the acute origin of a diaphragm paralysis patients get suddenly severely impaired which is interfering enormously with their lives. As this is often happening in middle aged patients they often have to discontinue professional activities. This means that the potential impact of this disorder is huge from patient and societal perspective and needs to be assessed.

As both therapies are completely different for invasiveness, the investigators need to compare the side effects and possible complications. Possible complications of the surgery are infection, bleeding and abdominal pain while the well know side effects of ventilatory support are leakage of the mask, aerophagia and a-synchrony between breathing pattern of the patient and the ventilator. As this is also an important outcome of this pilot study participants will be closely monitored from the start of therapy and there will be a telephone call after 2 months

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* diagnosed with a unilateral diaphragm paralysis based on isolated phrenic nerve injury.

Unilateral diaphragm paralysis is defined as follows: complaints of dyspnea and / or orthopnea combined with a drop in VC of more than 15% when change from upright to supine position and a positive sniff test during fluoroscopy or ultrasonography. A positive sniff test means that the diaphragm stands still or even moves in cranial direction (paradoxical movement ) during the sniff inspiratory maneuver.

* Ability to provide written consent
* Time between diagnosis and treatment should be at least 1 year

Exclusion Criteria:

* Patients diagnosed with a bilateral diaphragm paralysis.
* A diaphragm paralysis in combination with a more systemic neurological or neuromuscular disorder like for example Amyotrophic Lateral Sclerosis ,
* Hypercapnia during daytime (PaCO2 > 6.0 kPa)
* Radiotherapy of the thorax
* Contra indication for diaphragm surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparing surgical plication versus non-invasive ventilation . | 0-15 months
  10 patients surgical plication and 10 patients non-invasive ventilation while on the waiting list
Change in EuorQOL 5 Dimensions 5 Level (EQ-5D-5L questionnaire) range 1-1-1-1-1 (best score) to 5-5-5-5-5 (worst score) | baseline and 3 and 6 months
  questionnaire to score QUALY

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wijkstra, prof, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No